CLINICAL TRIAL: NCT04406272
Title: A Randomized, Controlled Phase II Surgical Trial to Evaluate Early Immunologic Pharmacodynamic Parameters for the Viral Cancer Therapy Ofranergene Obadenovec (VB-111) in Patients With Surgically Accessible Recurrent/Progressive Glioblastoma
Brief Title: VB-111 in Surgically Accessible Recurrent/Progressive GBM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial stopped at request of VBL Therapeutics, as they are no longer pursuing their VB-111 development program.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Principal Investigator, Patrick Wen, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-792
Record Dates: First submitted 2020-05-15; First posted 2020-05-28 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Recurrent Glioblastoma
Keywords: Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Surgical Procedures, Operative; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Before and After Surgery (Experimental): VB-111 will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovering from surgery (within 28-35 days after surgery), participants will receive intravenous VB-111 every 6 weeks. Participants evidencing disease progression may initiate bevacizumab at a pre-determined dose as needed for supportive care and will continue with VB-111 infusions every 6 weeks until tumor growth is evidenced a two consecutive time points.
  Interventions: Drug: VB11; Procedure: Surgery; Drug: Bevacizumab
- After Surgery (Experimental): Placebo (IV solution with no medicine) will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovering from surgery (within 28-35 days after surgery), participants will receive intravenous VB-111 every 6 weeks. Participants evidencing disease progression may initiate bevacizumab at a pre-determined dose as needed for supportive care and will continue with VB-111 infusions every 6 weeks until tumor growth is evidenced a two consecutive time points.
  Interventions: Drug: VB11; Procedure: Surgery; Other: Placebo; Drug: Bevacizumab
- After Surgery Standard of Care (Experimental): Placebo (IV solution with no medicine) will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovery from surgery, participants will receive standard of care treatment every 6 weeks until tumor growth is evidenced a two consecutive time points.
  Interventions: Procedure: Surgery; Other: Placebo

INTERVENTIONS:
Drug: VB11 — Intravenously administered type of gene therapy that works by blocking the process of blood-vessel creation. Disrupting a cancer from growing blood vessels, might slow the growth of the cancer or shrink it.
  Other Names: Ofranergene obadenovec
  Arms: After Surgery; Before and After Surgery
Procedure: Surgery — Treatment of disease or injury by cutting, abrading, suturing, or otherwise physically changing body tissues and organs.
Other: Placebo — Intravenous solution that has no therapeutic effect, used as a control in testing investigational drug.
  Arms: After Surgery; After Surgery Standard of Care
Drug: Bevacizumab — A type of antibody, Bevacizumab is intravenously administered and works by binding to and disrupting the vascular endothelial growth factor (VEGF). VEGF is a signal protein produced by cells that stimulates the formation of blood vessels. By disrupting VEGF, Bevacizumab helps to prevent the growth and maintenance of tumor blood vessels.
  Other Names: Avastin
  Arms: After Surgery; Before and After Surgery

SUMMARY:
This research study is studying a new viral cancer therapy, ofranergene obadenovec (VB-111), for recurrent or progressive glioblastoma (GBM), a brain tumor that is growing or progressing despite earlier treatment.

DETAILED DESCRIPTION:
This is a randomized, controlled, blinded, phase II, surgical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether it works in treating a specific disease. "Investigational" means that the drug is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved this intervention for recurrent or progressive glioblastoma.

In this research study, ofranergene obadenovec (VB-111) is the investigational drug being studied. VB-111 has been studied in lab experiments and in other types of cancer, and information from these studies suggest that it may be beneficial for recurrent or progressive glioblastoma.

VB-111 works by targeting and damaging the blood vessels that grow and nourish cancerous tumors leading to tumor starvation.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. After enrollment, participants will be randomized into one of three study groups. Randomization means that participants are put into a group by chance. Neither the participant nor the research doctor will choose what group a participant will be in.

* In group A participants receive VB-111 before and after surgery.
* In group B participants receive VB-111 after surgery.
* In group C participants won't receive VB-111 but would receive standard of care.

Treatment will be provided blindly, meaning participants do not know (are blinded as to) what treatment they are receiving to ensure that the results are not affected by a placebo effect (the power of suggestion). Participants will be given a study medication and it will contain either VB-111 or placebo (IV solution with no medicine).

VBL Therapeutics is supporting this research study by providing funding for the research study and the study drug.

Participants will be in this research study for as long as they do not have serious side effects and their disease does not get worse. It is expected that about 45 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria: ° ± µ ™ ®

* Histologically confirmed World Health Organization Grade IV malignant glioma (glioblastoma or gliosarcoma).
* First or second progression of glioblastoma/gliosarcoma (according to RANO criteria) following standard of care treatment upon initial diagnosis with radiation.
* Measurable disease by RANO criteria at progression.
* The maximal tumor volume at baseline meets the following criteria as determined by a local site investigator or surgeon: Longest diameter ≤ 4CM.
* Surgically resectable disease at progression.
* An interval of the following durations prior to randomization:

  * At least 28 days from prior surgical resection, or 7 days from stereotactic biopsy
  * At least 12 weeks from prior radiotherapy, unless there is unequivocal histologic confirmation of tumor progression
  * At least 23 days from prior chemotherapy
  * At least 42 days from nitrosureas
  * At least 42 days from other anti-tumor therapies (including vaccines)
  * At least 28 days from any investigational agent NOTE: no wash-out period required from TTF.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (including but not limited to exceptions of alopecia, laboratory values listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide.
* Corticosteroid use at or less than dexamethasone 2mg daily. Participants should be on a stable or decreasing dose for at least 7 days prior to randomization.
* Age ≥ 18 years on day of signing informed consent
* KPS ≥ 70% (see Appendix A)
* Adequate bone marrow, liver, and renal function according to the following criteria:

  * Absolute neutrophil count ≥ 1,500 cells/mL ~ 1.5 K/μL
  * Platelets ≥ 100,000 cells/mL ~ 100 K/μL
  * Total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for subjects with total bilirubin levels > 1.5 institutional ULN
  * Aspartate aminotransferase (AST) ≤ 2.0 x ULN
  * Serum creatinine level ≤ ULN or creatinine clearance ≥ 50 mL/min for participants with creatinine levels above normal limits (calculated by the Cockcroft-Gault formula)
* Ability to understand and willingness to sign a written informed consent document
* Availability of 10 unstained formalin-fixed paraffin-embedded slides.
* MRI within 14 days prior to registration.

  * NOTE: Due to the fact that the screening MRI will not be used for response purpose, participants may be registered if screening CT or MRI is > 14 days of registration if prospective approval is received from Overall PI
* Women of childbearing potential must have a negative serum beta-human chorionic gonadotropin urine or serum pregnancy test within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * NOTE: Women are considered postmenopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (withor without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment if she is considered not of child bearing potential.
* Males and females of childbearing potential must utilize a standard contraception method throughout the trial and up to 120 days after the last dose of treatment on study.

  * NOTE: Women of childbearing potential and men with female spouses of childbearing potential must agree to use two methods of reliable contraception simultaneously or to practice complete abstinence from heterosexual contact prior to study entry, while receiving treatment, and for 4 months after undergoing treatment. One method must include a highly effective method such as an intrauterine device, hormonal (birth control pills, injections or implants), tubal ligation or partner's vasectomy. The other method can be an additional hormonal therapy or barrier method such as a male condom, diaphragm or cervical cap. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in the study, she should inform her treating physician immediately

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has tumor primarily localized to the brainstem or spinal cord
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment
* Minor surgical procedure (e.g. stereotactic biopsy or shunt placement) within 7 days of first study treatment, placement of vascular access within 2 days of first study treatment
* Expected to have surgery other than the neurosurgical procedure intended for the GBM lesion during study treatment period
* Prior stereotactic radiotherapy (Note: those who have had biopsy proven tumor recurrence at a site of SRS treatment should be considered eligible if approved by the study central Investigator)
* Prior anti-angiogenic therapy including VEGF sequestering agents (i.e. bevacizumab, aflibercept, etc.) or VEGFR inhibitors (cedirinib, pazopanib, sunitinib, sorafenib, etc.)
* Prior administration of the study drug VB-111
* Concomitant medication that may interfere with study results (e.g. immunosuppressive agents other than inhaled, topical or intra-articular steroids or a stable or decreasing dose of oral corticosteroids of up to <2 mg/day dexamethasone equivalent)
* Known active second malignancy. Exceptions include non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast. Participants are not considered to have currently active malignancy if they have completed anticancer therapy and have been disease free for greater than 2 years prior to screening
* Uncontrolled intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of stroke or transient ischemic attack within 6 months prior to randomization
* Evidence of CNS hemorrhage CTCAE grade 2 or above on screening MRI
* Active cardiac disease within 6 months prior to randomization (i.e. acute coronary syndrome, unstable angina, New York Heart Association grade II or greater congestive heart failure, or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment)
* Significant vascular disease within 6 months prior to randomization (e.g. aortic aneurysm requiring surgical repair, peripheral arterial thrombosis, symptomatic peripheral vascular disease)
* History of venous thromboembolism CTCAE version 5.0 grade 3 or greater
* Known proliferative and/or vascular retinopathy
* Inadequately controlled hypertension (defined as systolic blood pressure > 150mmHg and/or diastolic blood pressure > 100mmHg) within 1 week of randomization
* History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 6 months of randomization.
* History of active gastrointestinal bleeding within 6 months prior to randomization.
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e. in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study randomization) use of aspirin > 325mg/day, clopidogrel > 75mg/day or equivalent. Therapeutic or prophylactic use of anticoagulants is allowed
* Known liver disease (alcoholic, drug/toxin induced, genetic or autoimmune)
* History of gastrointestinal perforation or abscess
* Positive testing to any of the following viruses: HIV, HBV, HCV within the last 6 months. Exceptions include participants with serology positive for HBV indicating past exposure but without evidence of active infection (e.g. negative PCR)
* History of intracranial abscess within 6 months prior to randomization
* Serious non-healing wound, active ulcer, or untreated bone fracture
* Pregnant or breastfeeding participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UT Health San Antonio MD Anderson Cancer Center (Mays Cancer Center), San Antonio, Texas
  - Huntsman Cancer Institute (HCI), University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: VB-111 Before and After Surgery: VB-111 will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovering from surgery (within 28-35 days after surgery), participants will receive intravenous VB-111 every 6 weeks. Participants evidencing disease progression may initiate bevacizumab at a pre-determined dose as needed for supportive care and will continue with VB-111 infusions every 6 weeks until tumor growth is evidenced a two consecutive time points.
  VB11: Intravenously administered type of gene therapy that works by blocking the process of blood-vessel creation. Disrupting a cancer from growing blood vessels, might slow the growth of the cancer or shrink it.
  Surgery: Treatment of disease or injury by cutting, abrading, suturing, or otherwise physically changing body tissues and organs.
  Bevacizumab: A type of antibody, Bevacizumab is intravenously administered and works by binding to and disrupting the vascular endothelial growth factor (VEGF). VEGF is a signal protein produced by cells that stimulates the formation of blood vessels. By disrupting VEGF, Bevacizumab helps to prevent the growth and maintenance of tumor blood vessels.
- Group B: Placebo Before Surgery; VB-111 After Surgery: Placebo (IV solution with no medicine) will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovering from surgery (within 28-35 days after surgery), participants will receive intravenous VB-111 every 6 weeks. Participants evidencing disease progression may initiate bevacizumab at a pre-determined dose as needed for supportive care and will continue with VB-111 infusions every 6 weeks until tumor growth is evidenced a two consecutive time points.
  VB11: Intravenously administered type of gene therapy that works by blocking the process of blood-vessel creation. Disrupting a cancer from growing blood vessels, might slow the growth of the cancer or shrink it.
  Surgery: Treatment of disease or injury by cutting, abrading, suturing, or otherwise physically changing body tissues and organs.
  Placebo: Intravenous solution that has no therapeutic effect, used as a control in testing investigational drug.
  Bevacizumab: A type of antibody, Bevacizumab is intravenously administered and works by binding to and disrupting the vascular endothelial growth factor (VEGF). VEGF is a signal protein produced by cells that stimulates the formation of blood vessels. By disrupting VEGF, Bevacizumab helps to prevent the growth and maintenance of tumor blood vessels.
- Group C: Placebo Before Surgery; Standard of Care After Surgery: Placebo (IV solution with no medicine) will be administered intravenously at a pre-determined dose at 14-28 days prior to surgery.
  Upon recovery from surgery, participants will receive standard of care treatment every 6 weeks until tumor growth is evidenced a two consecutive time points.
  Surgery: Treatment of disease or injury by cutting, abrading, suturing, or otherwise physically changing body tissues and organs.
  Placebo: Intravenous solution that has no therapeutic effect, used as a control in testing investigational drug.
Period: NeoAdjuvant Treatment
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Started | 6 | 4 | 5
Completed | 6 | 4 | 5
Not Completed | 0 | 0 | 0
Period: Adjuvant Therapy (Post-surgical)
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Started | 5 (One Group A subject withdrew consent to continue on active study treatment after surgery but prior to initiating any adjuvant therapy.) | 4 | 5
Completed | 5 | 4 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery | Total
Number analyzed (Participants) | 6 | 4 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 11
  >=65 years | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 4 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 4 | 1 | 3 | 8
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 2 | 4 | 12
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 2
Baseline Tumor Size [Count of Participants; unit: Participants]
  </= 15 cc | 4 | 3 | 2 | 9
  > 15 cc | 2 | 1 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Tumor Infiltrating T Cell (TIL) Density
Description: TIL Density Analysis was not - and will not be - performed on study samples, therefore no data was generated for this study objective.
  * Tumor infiltrating T cell (TIL) density is defined as the number of T lymphocytes per nucleated cell, and calculated by detailed sequencing of recombined T cell receptor sequences obtained from the tumor specimen gDNA.
  * Plan had been to use a two-sample t-test with tumor size stratification to test the difference of tumor infiltrating T cell density between the two groups (Group A vs combined Group B+C).
Time Frame: 2 years
Population: TIL Density Analysis was not - and will not be - performed on study samples, therefore no data was generated for this study objective. Because the trial was stopped after accrual of only 15 of 45 planned patients, it is believed that any results generated would not be of value, as there is no meaningful correlation that could be be drawn.
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: # of Participants to Experience a Reportable SAE on Study
Description: AEs graded using CTCAE version 5.0 criteria. Safety will be assessed by quantifying the toxicities and grades experienced by participants who have received VB-111, including serious adverse events (SAEs) All participants who receive at least one dose of VB-111/placebo will be evaluable for toxicity from the time of their first treatment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Number analyzed (Participants) | 6 | 4 | 5
Participants | 3 | 1 | 2

3. Secondary Outcome: 6-month Progression-free Survival (PFS-6)
Description: Defined as the %age of participants with progression-free survival at 6 months from surgery as defined by RANO. Recurrent/progressive GBM participants treated with VB-111 (Group A and Group B) compared to control (Group C), using RANO criteria. Progression is defined using Radiologic Assessment in Neuro-Oncology (RANO) criteria, as any of the following:
  * ≥ 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement, on stable or increasing doses of corticosteroids
  * Any new lesion
  * Significant increase in T2/FLAIR non-enhancing lesions on stable or increasing doses of corticosteroids not felt to be caused by co-morbid events
  * Clear clinical deterioration not attributable to other causes apart from the tumor or changes in corticosteroid dose
  * Clear progression of non-measurable disease
  * Or failure to return for evaluation due to death or deteriorating condition
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Number analyzed (Participants) | 6 | 4 | 5
Participants | 1 | 1 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS, analyses will be conducted using historical comparison data which are available from a pooled analysis of Phase II experience in recurrent Grade IV gliomas who have undergone surgery either just prior to starting treatment or as part of. Kaplan-Meier (KM) curves and median estimates from the KM curves will be provided as appropriate. Participants without efficacy evaluation data or without survival data will be censored at Day 1. For evaluation of the expansion of TCR clones, a two-sample T-test with Bonferroni adjustment will be used to compare the increase number of expanded TCR clones after VB-111 in Group A+B vs Group C.
Time Frame: Time from randomization until death from any cause; 37 months was the maximum time a participant remained in follow-up before passing away (10 pts), withdrawing consent (2 pts), being lost to follow-up (2 pts), or trial termination (1 pt).
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
Number analyzed (Participants) | 6 | 4 | 5
Participants
  <5 months | 2 | 1 | 0
  6-10 months | 3 | 1 | 2
  11-15 months | 0 | 1 | 1
  16-20 months | 0 | 0 | 2
  > 20 months | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) monitored/assessed up to 2 years (as the maximum # of days a patient was on active study treatment was 665 days). AEs are collected from the time of screening through 30 days following end of study treatment and any AEs meeting serious criteria through 90 days following end of study treatment.
Description: An AE is any undesirable sign, symptom or medical condition that develops or worsens in severity after initiating study treatment or any protocol-specified procedure, regardless of attribution. An SAE is any AE at any dose & regardless of causality that: results in death, is life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is an important medical event.
Arm/Group | Group A: VB-111 Before and After Surgery | Group B: Placebo Before Surgery; VB-111 After Surgery | Group C: Placebo Before Surgery; Standard of Care After Surgery
All-Cause Mortality (participants affected / at risk) | 3/6 | 2/4 | 5/5
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/4 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: VB-111 Before and After Surgery (N=6) | Group B: Placebo Before Surgery; VB-111 After Surgery (N=4) | Group C: Placebo Before Surgery; Standard of Care After Surgery (N=5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Memingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify: Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other, specify: Elevated WBC in CSF (Investigations) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Skin & subcutaneous tissue disorders - Other, specify: Preseptal cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: VB-111 Before and After Surgery (N=6) | Group B: Placebo Before Surgery; VB-111 After Surgery (N=4) | Group C: Placebo Before Surgery; Standard of Care After Surgery (N=5)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Ear & labyrinth disorders - Other, specify: right otitis media (Ear and labyrinth disorders) | 1 | 0 | 0
Eye disorders - Other, specify: Vision disorder - L quadrantopia (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Chills (General disorders) | 2 | 2 | 0
Edema limbs (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 4 | 1 | 2
Fever (General disorders) | 3 | 1 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0 | 0
Infections & infestations - Other, specify: COVID-19 (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 2 | 3 | 1
Platelet count decreased (Investigations) | 1 | 0 | 3
White blood cell decreased (Investigations) | 0 | 2 | 1
Investigations - Other, specify: Abdomen muscle pain (Investigations) | 0 | 0 | 1
Investigations - Other, specify: Knee muscle pain (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolism & nutrition disorders - Other, specify: Lactate level increased (Metabolism and nutrition disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 0 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 1
Memory impairment (Nervous system disorders) | 2 | 0 | 0
Muscle weakness left-sided (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 1
Nervous system disorders - Other, specify: Baseline pain in his bilateral lower extremities (Nervous system disorders) | 0 | 0 | 1
Nervous system disorders - Other, specify: Cognitive dysfunction (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2
Thromboembolic event (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT04406272/Prot_SAP_000.pdf